CLINICAL TRIAL: NCT06632054
Title: Use of Text Messaging Reminders to Increase FIT Completion Among Patients at the New York University (NYU) Family Health Centers (FHCs)
Brief Title: Use of Text Messaging Reminders to Increase FIT Completion Among Patients at the NYU FHCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QI- Fit Testing Trial
Record Dates: First submitted 2024-10-07; First posted 2024-10-08 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Text Message Reminders (Experimental): Participants will receive text message reminders to complete FIT for colon cancer screening.
  Interventions: Behavioral: Text Message Reminders
- Usual Care (Phone Call Reminders) (No Intervention): Participants will receive usual care (phone call reminders to complete FIT for colon cancer screening).

INTERVENTIONS:
Behavioral: Text Message Reminders — Text message reminders (instead of usual care - phone call reminders) to complete FIT for colon cancer screening.
  Arms: Text Message Reminders

SUMMARY:
The research team will compare the efficacy of targeted text message reminders against currently used phone call reminders at increasing patient completion of fecal immunochemical test (FIT) for colon cancer screening.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients eligible for FIT at a Family Health Center clinic (excluding Flatbush locations).

Exclusion Criteria:

* See inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1283 (Actual)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
FIT Completion at 7 Days Post-FIT Test Order | Day 7 Post-Visit
FIT Completion at 14 Days Post-FIT Test Order | Day 14 Post-Visit
FIT Completion at 21 Days Post-FIT Test Order | Day 21 Post-Visit

SECONDARY OUTCOMES:
Total Time to Completion of FIT Test | Up to Day 21 Post-Visit

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horwitz, MD, MHS, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a quality improvement (QI) project and individual participant data (IPD) will not be shared with other researchers.